CLINICAL TRIAL: NCT04121247
Title: Nonpharmacological Approaches Used by Parents of Children With Sickle Cell Disease and the Effectiveness of Education Given to Nonpharmacological Approaches
Brief Title: Nonpharmacological Approaches and Parental Education in Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Emine EFE, Prof.Dr., Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AkdenizUnursingfaculty
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Nursing Caries
Keywords: sickle cell disease; nonpharmacological approaches; pain; parent; nurse
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Intervention Model Description: the type of initiative tests to determine the effectiveness of education provided to parents in both countries.
  However, it tests the non-pharmacological approaches used by parents between the two countries.
Who Masked: Participant, Care Provider
Masking Description: parents and care provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Parents in Chad will be trained (Experimental): The education was given individually by the researcher (first researcher / author), before examining the child's doctor. The interactive education was completed in 30-40 min, using questions-answers. The education was conducted by the researcher using the education book.
  Interventions: Other: nonpharmacological approaches to parents of children with sickle cell disease training program
- Experimental: Parents in Turkey will be trained (Experimental): The education was given individually by the researcher (first researcher / author), before examining the child's doctor. The interactive education was completed in 30-40 min, using questions-answers. The education was conducted by the researcher using the education book.
  Interventions: Other: nonpharmacological approaches to parents of children with sickle cell disease training program

INTERVENTIONS:
Other: nonpharmacological approaches to parents of children with sickle cell disease training program — use of non-pharmacological approaches in children with sickle cell disease, parent education

SUMMARY:
Aim: Sickle cell disease (SCD) is a hereditary disease. Approximately 5% of the world's population carries trait genes for haemoglobin disorders, mainly, sickle-cell disease and thalassaemia. The incidence of sickle cell disease varies according to different geographical locations. Persons with SCD experience both acute and chronic pain. it is important that nonpharmacological therapies be investigated and used as complements to pharmacological therapies to address and treat both acute and chronic pain for those with SCD. An educational program involving parents with children with SCD can help parents use nonpharmacological methods for their children in reducing pain. The training program allows parents to develop their knowledge of the SCD and the importance of non-pharmacological methods, and may provide parents with the opportunity to develop preventive attitudes towards reducing pain crises. The research has two purposes. The first is to identify the non-pharmacological approaches that parents use to help their children with sickle cell disease in Turkey, Chad. Second, to determine the effectiveness of non-pharmacological approaches given to parents in Turkey, Chad.

Method: This study is an experimental research method using a quasi-experimental design. This study used a pretest and posttest, with a design that is used is the two group pretest-posttest design. The study was conducted on the parents of children with sickle cell disease diagnosed and followed up in the Pediatric Hematology Oncology polyclinics of two hospitals in Chad in Central Africa between September 2015 and February 2016. The study found in April 2016 and July 2016 between Turkey's southern Antalya and Mersin two university hospital outpatient Children's pediatric hematology oncology has made clinic on sickle cell disease diagnosed and monitored the children's parents. The parents were selected using eligibility criteria and the study was performed in three steps (Pre-intervention testing session, education session, and post-intervention testing session). In the first step, "Information Form", "Parents' Experience of Nonpharmacological Methods Questionnaire", and "Nonpharmacological Approaches Used by Parents for Their Children and Knowledge of Parents about Nonpharmacological Approaches Questionnaire" questionnaires were applied to parents. In the second step an individual education was conducted by the researcher using the education book. In the third step, the questionnaire were reapplied after 3 weeks.

DETAILED DESCRIPTION:
In this study, nonpharmacological approaches used by parents of sickle cell anemia patients were determined. However, the effectiveness of the education given to non-pharmacological approaches to parents was examined.

The study was first applied to parents in Chad. Then applied to parents in Turkey. n the study, parents' experience of nonpharmacological approaches questionnaire was used.

The form consisted of 8 multiple-choice questions, including a single open-ended question. If the parent used a nonpharmacological approach for the child, the name of the nonpharmacological approach (open - ended question) was written on the form.

In addition, the form was asked to write the frequency of using a nonpharmacological approach (sometimes / always / not use). Parents' pre- and post-educational knowledge of non-pharmacological methods to reduce the pain of children with SCD was measured with a closed-ended questionnaire developed by the researchers in the literature (he knows/he does not know). Nonpharmacological approaches in sickle cell disease training book was the intervention of this study. Nonpharmacological approaches in sickle cell disease training book "Parental Education Program for Nonpharmacological Approaches Used in Pain in Children with Sickle Cell Disease", was prepared according to previous studies by the researchers. The language used for administration of the instruments and the language used in education book was French / Arabic / Turkish.

ELIGIBILITY:
Inclusion Criteria:

* Turkish is spoken by parents and in Chad, parents can speak either Arabic or French
* that at least one member of the family knows how to either read or write
* parents agreeing to face-to-face interviewing

Exclusion Criteria:

* the participant to come out of his own accord

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-02 (Actual)

PRIMARY OUTCOMES:
Information form | In one week
  The information questionnaire contains information about parents and children. Parents; age, parents participating in the survey, education, occupation, marital status. Children; age, sex, number of siblings diagnosed with SCD, frequency of the child's pain crisis, medicines or drugs used by the child.
Parents' experience of nonpharmacological approaches questionnaire | In one week
  The form consisted of 8 multiple-choice questions, including the experience of parents using nonpharmacological approaches on SCD pain in their children, and asked for the name of the method using a single open-ended question. If the parent used nonpharmacological approach for the child, the name of the nonpharmacological approach (open-ended question) was written on the form.
  In addition, the form was asked to write the frequency of using nonpharmacological approach (sometimes/always/not use). The questionnaire about the nonpharmacological approach used by the parents was created by the researchers. This form, prepared by the researcher according to the literature, includes nonpharmacological approaches that parents can use in pain crisis.
Nonpharmacological approaches of pain relief parental information questionnaire | In three weeks
  Parents' pre- and post-educational knowledge of non-pharmacological methods to reduce the pain of children with SCD was measured with a closed-ended questionnaire developed by the researchers in the literature (he knows/he does not know).
  Nonpharmacological approaches of pain relief parental information questionnaire was prepared according to previous studies by the researchers (Williams&Tanabe, 2016; Wong, 2013; Demir, 2012; Monti&Yang, 2005; Delicou & Maragkos, 2013).
  Five expert opinions were consulted for the understandability of the questionnaire before the study. Two of them were doctors specializing in Sickle Cell Disease and three of them were the lecturers of the nursing department.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz University
Locations (1):
- Emine EFE, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date

REFERENCES:
- [Background] Crosby LE, Simmons K, Kaiser P, Davis B, Boyd P, Eichhorn T, Mahaney T, Joffe N, Morgan D, Schibler K, Anderson V, Quinn CT, Kalinyak KA. Using Quality Improvement Methods to Implement an Electronic Medical Record (EMR) Supported Individualized Home Pain Management Plan for Children with Sickle Cell Disease. J Clin Outcomes Manag. 2014 May;21(5):210-217. PMID 25258504
- [Background] Dampier C, Ely B, Brodecki D, Coleman C, Aertker L, Sendecki JA, Leiby B, Kesler K, Hyslop T, Stuart M. Pain characteristics and age-related pain trajectories in infants and young children with sickle cell disease. Pediatr Blood Cancer. 2014 Feb;61(2):291-6. doi: 10.1002/pbc.24796. Epub 2013 Sep 24. PMID 24115743
- [Background] Majumdar S, Thompson W, Ahmad N, Gordon C, Addison C. The use and effectiveness of complementary and alternative medicine for pain in sickle cell anemia. Complement Ther Clin Pract. 2013 Nov;19(4):184-7. doi: 10.1016/j.ctcp.2013.05.003. Epub 2013 Jun 22. PMID 24199970
- [Background] Makani J, Williams TN, Marsh K. Sickle cell disease in Africa: burden and research priorities. Ann Trop Med Parasitol. 2007 Jan;101(1):3-14. doi: 10.1179/136485907X154638. PMID 17244405
- [Background] Williams H, Tanabe P. Sickle Cell Disease: A Review of Nonpharmacological Approaches for Pain. J Pain Symptom Manage. 2016 Feb;51(2):163-77. doi: 10.1016/j.jpainsymman.2015.10.017. Epub 2015 Nov 17. PMID 26596876
- [Background] Thompson WE, Eriator I. Pain control in sickle cell disease patients: use of complementary and alternative medicine. Pain Med. 2014 Feb;15(2):241-6. doi: 10.1111/pme.12292. PMID 24524842
- [Background] Wilson BH, Nelson J. Sickle cell disease pain management in adolescents: a literature review. Pain Manag Nurs. 2015 Apr;16(2):146-51. doi: 10.1016/j.pmn.2014.05.015. Epub 2014 Aug 28. PMID 25175555
- [Background] Matthie N, Jenerette C. Understanding the Self-Management Practices of Young Adults with Sickle Cell Disease. J Sick Cell Dis Hemoglobinopathies. 2017 May;2017:76-87. PMID 30505880
- [Background] Ratanawongsa N, Haywood C Jr, Bediako SM, Lattimer L, Lanzkron S, Hill PM, Powe NR, Beach MC. Health care provider attitudes toward patients with acute vaso-occlusive crisis due to sickle cell disease: development of a scale. Patient Educ Couns. 2009 Aug;76(2):272-8. doi: 10.1016/j.pec.2009.01.007. Epub 2009 Feb 23. PMID 19233587